CLINICAL TRIAL: NCT05196386
Title: Usual Care Intervention Research Evaluating the Impact of a Personalized Pharmaceutical Plan on the Duration of Opioid Treatment in Non-cancerous Pain
Acronym: PPP-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/0025/HP
Record Dates: First submitted 2020-02-04; First posted 2022-01-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Non-cancerous Pain; Opioid Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with targeted pharmaceutical interview (Experimental): Specific information about treatment delivered by pharmacist
  Interventions: Behavioral: Admission conciliation interview; Behavioral: Discharge conciliation interview; Behavioral: Targeted pharmaceutical interview
- Patient without targeted pharmaceutical interview (Other): No Specific information about treatment delivered by pharmacist
  Interventions: Behavioral: Admission conciliation interview; Behavioral: Discharge conciliation interview

INTERVENTIONS:
Behavioral: Admission conciliation interview — Previous treatment conciliation at hospital admission
Behavioral: Discharge conciliation interview — Allocated treatment during hospital stay
Behavioral: Targeted pharmaceutical interview — Specific information about treatment delivered by pharmacist
  Arms: Patient with targeted pharmaceutical interview

SUMMARY:
Many treatments with WHO grade III opioids are being introduced in the rheumatology department for non-cancerous pain. The duration of this treatment prescribed at discharge is often uncontrolled and sometimes leads to significant addiction.

The team at the local pain center recommends an average duration of 28 days for this type of pain. There is a full-time pharmacy intern in the rheumatology department.

The aim of this work is to evaluate the impact of a targeted pharmaceutical interview on the duration of the morphine treatment initiated during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 75 years old when entering the rheumatology department
* Hospitalization in the rheumatology department
* Patient with acute non-traumatic musculoskeletal disease
* Patient not taking grade III opioid treatment
* Patient affiliated to a social security scheme
* Patient having read and understood the information letter and signed the consent form
* Patient present on a day which the pharmacy intern is present

Exclusion Criteria:

* Presence of cancer, fibromyalgia, already diagnosed at inclusion
* Patient does not understand French
* Patient with Current or past opioid addiction
* Person deprived of liberty by administrative or judicial decision

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Total duration of opioid treatment | 6 months

SECONDARY OUTCOMES:
Rate of patients exceeding 28 days of cumulative duration of treatment | 6 months
Rate of patients exceeding 90 days of cumulative duration of treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier VITTECOQ, Pr, Principal Investigator — University Hospital, Rouen; Remi VARIN, Pr, Principal Investigator — University Hospital, Rouen; Catherine CHENAILLER, Dr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France